CLINICAL TRIAL: NCT03559855
Title: Evaluation of High School-based Relationship Education: Center for Relationship Education
Brief Title: Evaluation of High School-based Relationship Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Denver (Other)
Responsible Party: Principal Investigator, Galena Rhoades, Research Associate Professor, University of Denver
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 977115
Record Dates: First submitted 2018-05-23; First posted 2018-06-18 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Responsible Sex
MeSH Terms: conditions — Safe Sex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Essentials (Experimental): The Real Essentials curriculum is delivered in class to students by the Center for Relationship Education staff. It consists of 5 to 6 hours of healthy relationship education.
  Interventions: Behavioral: Real Essentials
- Class as Usual (No Intervention): For the Class-as-Usual condition, there is no change in class content. Teachers offer what they typically offer.

INTERVENTIONS:
Behavioral: Real Essentials — The REAL Essentials curriculum is a healthy relationship education program for youth developed by the Center for Relationship Education.
  Arms: Real Essentials

SUMMARY:
This study is a randomized controlled trial testing the effectiveness of a program provided in Colorado high schools by the Center for Relationship Education based in Denver, Colorado. 14 schools are randomly assigned to either provide the Real Essentials curriculum as part of health or similar classes or teach these classes as usual. The study design includes surveys administered pre-program, post-program and at 6-month and 12-month follow ups. Primary study outcomes are increased knowledge of healthy relationships and reduced risky sexual behavior.

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled in designated classes at 14 participating high schools schools in Colorado

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1135 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Healthy Relationship Knowledge and Skills | Change from pre-program through 1 year
  This outcome is measured by self-report survey.
Risky Sexual Behavior | Change from pre-program through 1 year
  This outcome is measured by self-report survey.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Denver, Denver, Colorado, United States